CLINICAL TRIAL: NCT02534233
Title: Evaluation of Effect of CryoBalloon Focal Ablation System on Human Esophageal Epithelium
Acronym: ColdPlay2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00075654
Record Dates: First submitted 2015-08-19; First posted 2015-08-27 (Estimated); Results first posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Barrett's Esophagus; Esophageal Squamous Dysplasia; Esophageal Cancer
Keywords: barrett's esophagus with dysplasia; early esophageal cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms | interventions — Cryosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CryoBalloon ablation (Experimental): Patients having ablation of dysplastic tissue in esophagus.
  Interventions: Device: CryoBalloon

INTERVENTIONS:
Device: CryoBalloon — Esophageal tissue ablation with focal freezing using nitrous oxide via a single use balloon catheter
  Other Names: Cryoablation

SUMMARY:
Assess Cryoablation (CryoBalloon Ablation cryotherapy) for treatment of Dysplastic Barrett's Esophagus, Esophageal Squamous Dysplasia and early Esophageal Cancer. The cryoablation treatment will be offered as an alternative to standard ablation therapies such as Radiofrequency Ablation, Argon Plasma Coagulation and carbon dioxide Cryotherapy).

DETAILED DESCRIPTION:
Cryoablation (cryotherapy) is an established type of mucosal ablation for treatment of various conditions in the GI tract, including Barrett's esophagus and esophageal cancer. The purpose of this study is to assess the safety, feasibility and performance of cryoablation system (the C2 Focal Cryoablation Device in patients with BE and esophageal squamous dysplasia who need ablation therapy for clinical standard care. The new cryoablation treatment will be offered as an alternative to standard ablation therapies already in place (radiofrequency ablation, carbon dioxide cryotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Patients recommended for ablation of either Barrett's esophagus with dysplasia or esophageal squamous dysplasia, scheduled for upper endoscopy.

Exclusion Criteria:

* Patient unable to undergo endoscopy,
* Patients with visible esophageal mass.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2024-08 (Actual); Study Completion 2025-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Canto, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Canto MI, Shaheen NJ, Almario JA, Voltaggio L, Montgomery E, Lightdale CJ. Multifocal nitrous oxide cryoballoon ablation with or without EMR for treatment of neoplastic Barrett's esophagus (with video). Gastrointest Endosc. 2018 Sep;88(3):438-446.e2. doi: 10.1016/j.gie.2018.03.024. Epub 2018 Apr 5. PMID 29626424
- [Result] Canto MI, Abrams JA, Kunzli HT, Weusten B, Komatsu Y, Jobe BA, Lightdale CJ. Nitrous oxide cryotherapy for treatment of esophageal squamous cell neoplasia: initial multicenter international experience with a novel portable cryoballoon ablation system (with video). Gastrointest Endosc. 2018 Feb;87(2):574-581. doi: 10.1016/j.gie.2017.07.013. Epub 2017 Jul 16. PMID 28720474
- See also: Durability of Cryoballoon Ablation in Neoplastic Barrett's Esophagus — https://doi.org/10.1016/j.tige.2021.11.007

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who are clinical patients of the Principal Investigator or Co-investigators will be identified as eligible by prior pathology proven biopsies with either Barrett's esophagus with dysplasia or esophageal squamous cell dysplasia.
  Recruitment will occur primarily in the outpatient GI clinic but can also be a phone contact and follow-up study consent for review with informed consent call.
Pre-assignment Details: 5 subjects were determined ineligible with index endoscopy finding exclusions, strictures restricting therapeutic scope or invasive disease.
Period: Overall Study
Arm/Group | CryoBalloon Ablation
Started | 53
12 Month | 51
Completed | 51
Not Completed | 2
Not completed — 2 participants with protocol deviations didn't complete | 2

BASELINE CHARACTERISTICS:
Arm/Group | CryoBalloon Ablation
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants] — eligibility criteria is age 18 years or greater
  Participants
    <=18 years | 0
    Between 18 and 65 years | 14
    >=65 years | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 45
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 53
Likert 11 Point Pain Score (0 no pain-10 worst) [Mean (Inter-Quartile Range); unit: units on a scale] — The 11-point Likert scale represents a range of discomfort or pain from 0 (no pain) to 10 (extreme pain), which individuals indicate their level of discomfort or pain
  units on a scale | 0 [0 to 3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Eradication of Esophageal Dysplasia
Description: Evaluate histopathology of esophageal tissue for absence of Barrett's esophagus or squamous dysplasia after cryoablation treatments (assess for complete eradication of dysplasia).
Time Frame: 12 months
Population: 51 assessable adult patients with data collected at 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CryoBalloon Ablation
Number analyzed (Participants) | 51
Participants | 51

2. Primary Outcome: Treatment-related Adverse Events Assessed by Pain Scale
Description: Evaluate by patient questionnaire for pain on an 11-point scale. The 11-point Likert scale represents a range of discomfort or pain from 0 (no pain) to 10 (extreme pain), which individuals indicate their level of discomfort or pain. Higher score more discomfort.
  Each subject is evaluated for post-treatment pain after each cryoablation session. Subjects may have a different number of treatment sessions depending on the extent of disease.
Time Frame: 1 day post treatment (day 2), 1 week post treatment (day 8), and 1 month (day 31)
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | CryoBalloon Ablation
Number analyzed (Participants) | 51
units on a scale
  Likert Pain score at 1 day post each cryoablation treatment | 1 [0 to 3]
  Likert Pain score at 1 week post each cryoablation treatment | 0 [0 to 3]
  Likert Pain score at 1 month post each (day 31 post each cryoablation treatment | 0 [0 to 3]

3. Primary Outcome: Treatment-related Adverse Events Assessed by Stricture Rate
Description: Number of patients with esophageal strictures requiring dilation. Patients reporting dysphagia with solid food, with balloon dilations from index visit to 12 months.
Time Frame: Up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | CryoBalloon Ablation
Number analyzed (Participants) | 51
Participants | 6

4. Secondary Outcome: Number of Participants With Complete Eradication of Intestinal Metaplasia
Description: Evaluate histopathology of esophageal tissue for absence of Barrett's esophagus (intestinal metaplasia) after cryoablation
Time Frame: 12 months
Population: 41 of the 51 evaluable subjects had Barrett's esophagus (intestinal metaplasia) data collected at 12 months; this outcome measure does not apply to subjects with esophageal squamous dyplasia.
Measure: Count of Participants; unit: Participants
Arm/Group | CryoBalloon Ablation
Number analyzed (Participants) | 41
Participants | 35

ADVERSE EVENTS:
Time Frame: Post ablation treatment assessment day 1, 7 days, 30 days, and follow up endoscopies up to 12 months
Description: pain (0-10 Likert pain scale,) pain requiring narcotics, dysphagia (0-4 dysphagia score), bleeding, esophageal strictures requiring dilation.
Arm/Group | CryoBalloon Ablation
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 9/53
Other Adverse Events (participants affected / at risk) | 0/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CryoBalloon Ablation (N=53)
GI Bleeding (Gastrointestinal disorders) | 1 (1) — Post esophageal cryoablation treatment bleeding requiring treatment
post cryoablation treatment pain requiring narcotics (Gastrointestinal disorders) | 2 (2) — subjects reporting pain requiring narcotics for pain at or between 1, 7, or 30 day follow up calls.
Esophageal stricture requiring dilation (Gastrointestinal disorders) | 6 (6) — subject reporting 3 or 4 on dysphagia scale, unable to swallow semi solid or liquid food

LIMITATIONS AND CAVEATS:
Prospective single arm non-randomized trial, no control subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02534233/Prot_SAP_000.pdf